CLINICAL TRIAL: NCT02683239
Title: A Phase 3 Randomized, Double-blind, Multi-Dose, Placebo-Controlled Study to Evaluate the Long-Term Safety and the Efficacy of Fasinumab in Patients With Pain Due to Osteoarthritis of the Knee or Hip
Brief Title: Long-Term Safety and Efficacy Study of Fasinumab in Patients With Pain Due to Osteoarthritis (OA) of the Knee or Hip
Acronym: FACT LTS & OA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R475-PN-1523; 2015-003783-36 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-17 (Estimated); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis of the Knee or Hip
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fasinumab dosing regimen 1 (Experimental)
  Interventions: Drug: Fasinumab
- Fasinumab dosing regimen 2 (Experimental)
  Interventions: Drug: Fasinumab
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fasinumab — Participants will receive sub-cutaneous (SC) injections of fasinumab
  Other Names: REGN475
  Arms: Fasinumab dosing regimen 1; Fasinumab dosing regimen 2
Drug: Placebo — Participants will receive sub-cutaneous (SC) injections of matching placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to describe the safety and tolerability of fasinumab, including adverse events of special interest (AESIs), in patients with pain due to radiographically-confirmed OA of the knee or hip.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female ≥18 years of age at the screening visit
2. Clinical diagnosis of OA of the knee or hip based on the American College of Rheumatology criteria with radiologic evidence of OA (K-L score ≥2) for the index joint at the screening visit
3. Moderate to severe pain in the index joint defined as a Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) average pain subscale score of ≥4
4. A history of 12 weeks of analgesic use for OA of the knee or hip
5. History of regular use of analgesic medications for OA pain

Key Exclusion Criteria:

1. History or presence at the screening visit of non OA inflammatory joint disease
2. History or presence on imaging of arthropathy, stress fracture, recent stress fracture, neuropathic joint arthropathy, hip dislocation, knee dislocation, congenital hip dysplasia with degenerative joint disease, extensive subchondral cysts, evidence of bone fragmentation or collapse, or primary metastatic tumor with the exception of chondromas or pathologic fracture during the screening period
3. Signs or symptoms of carpal tunnel syndrome within 6 months of screening
4. Patient is not a candidate for MRI
5. Is scheduled for a joint replacement surgery to be performed during the study period
6. Systemic (i.e., oral or intramuscular) corticosteroids within 30 days prior to the screening visit.
7. History or presence at the screening visit of multiple sclerosis, autonomic neuropathy, diabetic neuropathy, or other peripheral neuropathy, including reflex sympathetic dystrophy
8. History or diagnosis of chronic autonomic failure syndrome including pure autonomic failure, multiple system atrophy
9. Pregnant or breast-feeding women
10. Women of childbearing potential who have a positive pregnancy test result or do not have their pregnancy test result at baseline

Note: Other protocol defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5331 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (146):
- United States (50):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Investigational Site #1, Chandler, Arizona
  - Regeneron Investigational Site #2, Chandler, Arizona
  - Regeneron Investigational Site, Glendale, Arizona
  - Regeneron Investigational Site, Mesa, Arizona
  - Regeneron Investigational Site (4 locations), Phoenix, Arizona
  - Regeneron Investigational Site, Tempe, Arizona
  - Regeneron Investigational Site (2 locations), Tucson, Arizona
  - Regeneron Investigational Site, Little Rock, Arkansas
  - Regeneron Investigational Site, Beverly Hills, California
  - Regeneron Investigational Site, Carlsbad, California
  - Regeneron Investigational Site, San Diego, California
  - Regeneron Investigational Site, San Marcos, California
  - Regeneron Investigational Site, Vista, California
  - Regeneron Investigational Site, Aurora, Colorado
  - Regeneron Investigational Site, Colorado Springs, Colorado
  - Regeneron Investigational Site, Golden, Colorado
  - Regeneron Investigational Site, Littleton, Colorado
  - Regeneron Investigational Site, Clearwater, Florida
  - Regeneron Investigational Site, Orlando, Florida
  - Regeneron Investigational Site, Pinellas Park, Florida
  - Regeneron Investigational Site, Atlanta, Georgia
  - Regeneron Investigational Site (3 locations), Chicago, Illinois
  - Regeneron Investigational Site, Evansville, Illinois
  - Regeneron Investigational Site, Kansas City, Kansas
  - Regeneron Investigational Site, Frederick, Maryland
  - Regeneron Investigational Site, Worcester, Massachusetts
  - Regeneron Investigational Site, Richfield, Minnesota
  - Regeneron Investigational Site #1, St Louis, Missouri
  - Regeneron Investigational Site #2, St Louis, Missouri
  - Regeneron Investigational Site, Elkhorn, Nebraska
  - Regeneron Investigational Site, Fremont, Nebraska
  - Regeneron Investigational Site, Omaha, Nebraska
  - Regeneron Investigational Site, Las Vegas, Nevada
  - Regeneron Investigational Site, Jamaica, New York
  - Regeneron Investigational Site, New York, New York
  - Regeneron Investigational Site, High Point, North Carolina
  - Regeneron Investigational Site, Akron, Ohio
  - Regeneron Investigational Site, Cincinnati, Ohio
  - Regeneron Investigational Site, Columbus, Ohio
  - Regeneron Investigational Site, Oklahoma City, Oklahoma
  - Regeneron Investigational Site, Duncansville, Pennsylvania
  - Regeneron Investigational Site, Anderson, South Carolina
  - Regeneron Investigational Site, Greer, South Carolina
  - Regeneron Investigational Site #1, Dallas, Texas
  - Regeneron Investigational Site #2, Dallas, Texas
  - Regeneron Investigational Site, Houston, Texas
  - Regeneron Investigational Site, Lubbock, Texas
  - Regeneron Investigational Site, Plano, Texas
  - Regeneron Investigational Site, San Antonio, Texas
- Bulgaria (7):
  - Regeneron Investigational Site, Burgas
  - Regeneron Investigational Site #1, Plovdiv
  - Regeneron Investigational Site #2, Plovdiv
  - Regeneron Investigational Site #3, Plovdiv
  - Regeneron Investigational Site #1, Sofia
  - Regeneron Investigational Site #2, Sofia
  - Regeneron Investigational Site, Stara Zagora
- Regeneron Investigational Site, Santiago, Chile
- Colombia (2):
  - Regeneron Investigational Site, Bogotá
  - Regeneron Investigational Site, Medellín
- Denmark (3):
  - Regeneron Investigational Site, Aalborg
  - Regeneron Investigational Site, Ballerup Municipality
  - Regeneron Investigational Site, Vejle
- Estonia (2):
  - Regeneron Investigational Site, Paide
  - Regeneron Investigational Site, Tallinn
- Germany (5):
  - Regeneron Investigational Site, Leipzig, Saxony
  - Regeneron Investigational Site, Berlin
  - Regeneron Investigational Sites, Bochum
  - Regeneron Investigational Site, Frankfurt
  - Regeneron Investigational Site, Magdeburg
- Regeneron Investigational Site, Central, Hong Kong
- Hungary (5):
  - Regeneron Investigational Site, Budapest
  - Regeneron Investigational Site, Debrecen
  - Regeneron Investigational Site, Gyula
  - Regeneron Investigational Site, Hatvan
  - Regeneron Investigational Site, Zalaegerszeg
- Italy (2):
  - Regeneron Investigational Site, Florence
  - Regeneron Investigational Site, Naples
- Lithuania (4):
  - Regeneron Investigational Site, Alytus
  - Regeneron Investigational Site, Kaunas
  - Regeneron Investigational Site, Šiauliai
  - Regeneron Investigational Site, Vilnius
- Mexico (8):
  - Regeneron Investigational Site, Mexicali, Baja Californina
  - Regeneron Investigational Site, Guadalajara, Jalisco
  - Regeneron Investigational Site, Cuauhtémoc, Mexico City
  - Regeneron Investigational Site, Distrito Federal, Mexico City
  - Regeneron Investigational Site, Mexico City, Mexico City
  - Regeneron Investigational Site, Cuernavaca, Morelos
  - Regeneron Investigational Site, Culiacán, Sinaloa
  - Regeneron Investigational Site, Mérida, Yucatán
- Regeneron Investigational Site, Lima, Peru
- Poland (9):
  - Regeneron Investigational Site, Gdansk
  - Regeneron Investigational Site, Gdynia
  - Regeneron Investigational Site, Katowice
  - Regeneron Investigational Site, Krakow
  - Regeneron Investigational Site, Lodz
  - Regeneron Investigational Site, Poznan
  - Regeneron Investigational Site #1, Warsaw
  - Regeneron Investigational Site #2, Warsaw
  - Regeneron Investigational Site, Wroclaw
- Romania (2):
  - Regeneron Investigational Site #2, Bucharest
  - Regeneron Investigational Site #1, Bucharest
- Russia (6):
  - Regeneron Investigational Site, Kazan'
  - Regeneron Investigational Site, Novosibirsk
  - Regeneron Investigational Site, Samara
  - Regeneron Investigational Site, Tomsk
  - Regeneron Investigational Site #2, Yaroslavl
  - Regeneron Investigational Site #1, Yaroslavl
- South Africa (11):
  - Regeneron Investigational Site #1, Pretoria, Gauteng
  - Regeneron Investigational Site #2, Pretoria, Gauteng
  - Regeneron Investigational Site, Bloemfontein
  - Regeneron Investigational Site, Cape Town
  - Regeneron Investigational Site, Kempton Park
  - Regeneron Investigational Site, Parow
  - Regeneron Investigational Site, Port Elizabeth
  - Regeneron Investigational Site, Pretoria
  - Regeneron Investigational Site, Roodepoort
  - Regeneron Investigational Site, Somerset West
  - Regeneron Investigational Site, Soweto
- Spain (4):
  - Regeneron Investigational Site, A Coruña
  - Regeneron Investigational Site, Barcelona
  - Regeneron Investigational Site, Madrid
  - Regeneron Investigational Site, Seville
- Sweden (8):
  - Regeneron Investigational Site, Malmo, Skåne County
  - Regeneron Investigational Site, Borås
  - Regeneron Investigational Site, Gothenburg
  - Regeneron Investigational Site, Helsingborg
  - Regeneron Investigational Site, Linköping
  - Regeneron Investigational Site, Lund
  - Regeneron Investigational Site, Uppsala
  - Regeneron Investigational Site, Vällingby
- Ukraine (5):
  - Regeneron Investigational Site, Cherkasy
  - Regeneron Investigational Site #3, Kyiv
  - Regeneron Investigational Site #1, Kyiv
  - Regeneron Investigational Site #2, Kyiv
  - Regeneron Investigational Site, Lviv
- United Kingdom (10):
  - Regeneron Investigational Site, Birmingham
  - Regeneron Investigational Site, Chorley
  - Regeneron Investigational Site, Glasgow
  - Regeneron Investigational Site, Hexham
  - Regeneron Investigational Site, Liverpool
  - Regeneron Investigational Site, Manchester
  - Regeneron Investigational Site, Middlesex
  - Regeneron Investigational Site, Reading
  - Regeneron Investigational Site, Romford
  - Regeneron Investigational Site, Sidcup

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13,945 participants were screened. Of those, 5,331 met the eligibility criteria and were randomized to 1 of 7 treatment arms.
Groups:
- Fasinumab-matching Placebo Q4W/Q8W: Participants received fasinumab matching placebo SC injection, Q4W or Q8W from Day 1 up to 52 weeks.
- Fasinumab 1 mg SC Q8W: Participants received fasinumab 1 mg SC injection, Q8W from day 1 up to 52 weeks.
- Fasinumab 1 mg SC Q4W: Participants received fasinumab 1 mg SC injection Q4W from day 1 up to 52 weeks.
- Fasinumab 3 mg SC Q4W: Participants received fasinumab 3 mg SC injection, Q4W from day 1 up to 52 weeks.
- Fasinumab 6 mg SC Q8W: Participants received fasinumab 6 mg SC injection, Q8W from day 1 up to 52 weeks.
- Fasinumab 6 mg SC Q4W: Participants received fasinumab 6 mg SC injection Q4W from day 1 up to 37 weeks of 52-week treatment period.
- Fasinumab 9 mg SC Q4W: Participants received fasinumab 9 mg SC injection, Q4W from day 1 up to 37 weeks of 52-week treatment period.
Period: Overall Study
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Started | 1260 | 971 | 975 | 214 | 1680 | 116 | 115
Completed | 800 | 738 | 756 | 94 | 935 | 56 | 44
Not Completed | 460 | 233 | 219 | 120 | 745 | 60 | 71
Not completed — Protocol Violation | 35 | 23 | 26 | 4 | 35 | 4 | 5
Not completed — Adverse Event | 64 | 39 | 42 | 16 | 189 | 9 | 9
Not completed — Physician Decision | 38 | 19 | 14 | 73 | 143 | 14 | 15
Not completed — Withdrawal by Subject | 187 | 99 | 91 | 18 | 248 | 22 | 28
Not completed — Lost to Follow-up | 77 | 24 | 25 | 7 | 88 | 8 | 11
Not completed — Death | 9 | 5 | 8 | 0 | 12 | 1 | 0
Not completed — Lack of Efficacy | 50 | 23 | 12 | 2 | 29 | 2 | 3
Not completed — Missing data | 0 | 1 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set for the evaluation of long-term safety (FAS-LTS) included all randomized participants in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W | Total
Number analyzed (Participants) | 1260 | 971 | 975 | 214 | 1680 | 116 | 115 | 5331
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (9.24) | 65.0 (9.24) | 65.1 (8.57) | 65.3 (9.19) | 62.9 (9.61) | 62.4 (8.38) | 63.4 (9.89) | 64.0 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 913 | 723 | 705 | 149 | 1237 | 83 | 76 | 3886
  Male | 347 | 248 | 270 | 65 | 443 | 33 | 39 | 1445
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 117 | 177 | 182 | 6 | 124 | 8 | 8 | 622
  Not Hispanic or Latino | 1139 | 791 | 787 | 207 | 1547 | 108 | 107 | 4686
  Unknown or Not Reported | 4 | 3 | 6 | 1 | 9 | 0 | 0 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 50 | 53 | 0 | 8 | 0 | 1 | 131
  Asian | 25 | 7 | 9 | 0 | 52 | 0 | 0 | 93
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Black or African American | 156 | 64 | 66 | 16 | 213 | 15 | 12 | 542
  White | 996 | 759 | 738 | 190 | 1352 | 99 | 102 | 4236
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 63 | 91 | 109 | 8 | 55 | 1 | 0 | 327
Western Ontario and McMaster Universities Index of Osteoarthritis (WOMAC) Pain Subscale Score [Mean (Standard Deviation); unit: Score on a Scale] — The WOMAC index is comprised of 24 parameters grouped in 3 subscales (pain-5 questions, physical function -17 questions and stiffness - 2 questions), with 0-10 grading of each question. The scores for each subscale are summed up, divided by number of questions, and each subscale is reported using Numerical Rating Scale score of 0-10. In addition to subscales, a total score is provided as the sum of normalized subscale scores divided by three, and reported using a Numerical Rating Scale score of 0-10. Higher scores indicate worse pain, stiffness and functional limitations. Population: Baseline WOMAC score data were collected for index joint and only for participants in the sub-study.
  Score on a Scale
    number analyzed (Participants) | 214 | 214 | 217 | 213 | 213 | 0 | 0 | 1071
    (all) | 6.6 (1.55) | 6.70 (1.44) | 6.6 (1.49) | 6.5 (1.47) | 6.6 (1.41) |  |  | 6.6 (1.47)
WOMAC Physical Function Subscale Score [Mean (Standard Deviation); unit: Score on a Scale] — The WOMAC index is comprised of 24 parameters grouped in 3 subscales (pain-5 questions, physical function -17 questions and stiffness - 2 questions), with 0-10 grading of each question. The scores for each subscale are summed up, divided by number of questions, and each subscale is reported using Numerical Rating Scale score of 0-10. In addition to subscales, a total score is provided as the sum of normalized subscale scores divided by three, and reported using a Numerical Rating Scale score of 0-10. Higher scores indicate worse pain, stiffness and functional limitations. Population: Baseline WOMAC score data were collected for index joint and only for participants in the sub-study.
  Score on a Scale
    number analyzed (Participants) | 207 | 212 | 212 | 208 | 209 | 0 | 0 | 1048
    (all) | 6.47 (1.583) | 6.56 (1.631) | 6.41 (1.495) | 6.27 (1.699) | 6.38 (1.598) |  |  | 6.42 (1.602)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-Emergent Adverse Event (TEAE)
Time Frame: Baseline up to week 52
Population: The safety analysis set for the evaluation of long-term safety (SAF-LTS) included all randomized participants in the overall study who received any study drug; it was based on the treatment-as-received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants | 1055 | 840 | 885 | 185 | 1487 | 93 | 92

2. Primary Outcome: Number of Participants With Any Serious TEAE
Time Frame: Baseline up to week 52
Population: The SAF-LTS included all randomized participants in the overall study who received any study drug; it was based on the treatment-as-received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants | 82 | 57 | 70 | 13 | 107 | 5 | 3

3. Primary Outcome: Number of Participants With Any Adverse Event (AE) up to Week 72
Time Frame: Baseline up to week 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants | 1112 | 867 | 902 | 192 | 1570 | 106 | 106

4. Primary Outcome: Number of Participants With Any Serious AE up to Week 72
Time Frame: Baseline up to week 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants | 173 | 138 | 176 | 44 | 413 | 28 | 26

5. Primary Outcome: Number of Participants With Adjudicated Arthropathy (AA)
Description: Adjudicated arthropathy (AA) is a composite term that encompasses the following conditions: Rapidly progressive OA type 1 and 2, Subchondral insufficiency fractures, and Primary Osteonecrosis. AAs were also evaluated to determine if they met Destructive Arthropathy criteria.
Time Frame: Baseline up to week 52 and week 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants
  Week 52 | 23 | 52 | 62 | 25 | 238 | 14 | 8
  Week 72 | 32 | 71 | 89 | 27 | 303 | 18 | 13

6. Primary Outcome: Number of Participants With Adjudicated Arthropathy (AA) Meeting Destructive Arthropathy (DA) Criteria
Description: DA is a unique clinical form of rapidly destructive arthropathy over and above that seen in the normal progression of OA. DA criteria can be associated with Rapidly Progressive OA type 2, Subchondral Insufficiency fracture, and Primary Osteonecrosis confirmed by an arthropathy adjudication committee.
Time Frame: Baseline up to week 52 and week 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants
  Week 52 | 0 | 1 | 3 | 1 | 20 | 1 | 1
  Week 72 | 0 | 1 | 5 | 1 | 31 | 1 | 1

7. Primary Outcome: Number of Participants With at Least One Peripheral Sensory Event That Required a Neurology Consultation
Description: Any participant with a peripheral sensory event that persisted for 2 months was referred for a neurology or other specialty consultation and reported as an adverse event of special interest (AESI).
Time Frame: Baseline up to week 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants | 29 | 65 | 62 | 21 | 75 | 3 | 1

8. Primary Outcome: Number of Participants With Sympathetic Nervous System (SNS) Dysfunction
Description: Potential events of sympathetic nervous system (SNS) dysfunction were monitored throughout the study through physical examination, AE reporting, assessment of orthostatic hypotension, and the Survey of Autonomic Symptoms. Sympathetic nervous system dysfunction was diagnosed after consultation with an appropriate specialist, such as a neurologist and/or cardiologist.
Time Frame: Baseline up to week 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

9. Primary Outcome: Number of Participants With at Least One All-Cause Joint Replacement (JR) Surgery
Description: All joint replacement surgery events regardless of cause at weeks 52 and 72. An end of study phone contact was also conducted approximately 52 weeks following the last dose of study drug.
Time Frame: Baseline up to weeks 52, 72, and end of study (52 weeks post last dose)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants
  Week 52 | 37 | 27 | 37 | 15 | 109 | 8 | 4
  Week 72 | 55 | 55 | 71 | 23 | 197 | 11 | 9
  End of Study (52 weeks post-last dose) | 79 | 81 | 118 | 30 | 309 | 18 | 15

10. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Laboratory Values up to Week 52
Description: Number of participants with potentially clinically significant abnormal values in hematology, chemistry, and urinalysis during the treatment period were reported. Clinical significance was determined by the investigator.
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants
  Hematology: number analyzed (Participants) | 1016 | 854 | 875 | 176 | 1405 | 88 | 85
  Hematology | 195 | 236 | 241 | 28 | 304 | 7 | 11
  Chemistry: number analyzed (Participants) | 1181 | 941 | 950 | 207 | 1627 | 111 | 108
  Chemistry | 403 | 365 | 403 | 105 | 717 | 36 | 34
  Urinalysis: number analyzed (Participants) | 1131 | 940 | 949 | 207 | 1588 | 58 | 55
  Urinalysis | 32 | 42 | 45 | 2 | 55 | 1 | 1

11. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Laboratory Values Post-Treatment up to Week 72
Description: Number of participants with potentially clinically significant abnormal values in hematology, chemistry, and urinalysis during the post-treatment period were reported. Clinical significance was determined by the investigator.
Time Frame: End of treatment up to week 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1257 | 966 | 974 | 214 | 1677 | 116 | 115
Participants
  Hematology: number analyzed (Participants) | 1007 | 808 | 814 | 190 | 1426 | 104 | 100
  Hematology | 171 | 149 | 154 | 23 | 279 | 29 | 32
  Chemistry: number analyzed (Participants) | 1032 | 813 | 818 | 195 | 1459 | 107 | 100
  Chemistry | 267 | 228 | 225 | 59 | 474 | 36 | 40
  Urinalysis: number analyzed (Participants) | 1015 | 811 | 814 | 190 | 1442 | 103 | 99
  Urinalysis | 16 | 24 | 18 | 1 | 37 | 5 | 3

12. Primary Outcome: Number of Participants With Anti-drug Antibody (ADA) up to Week 72
Description: Immunogenicity was characterized by ADA responses & titers. Responses categories: Negative - ADA negative response at all time points, regardless of missing samples; Pre-existing immunoreactivity - ADA positive response at baseline with all post first dose negative results or positive response at baseline with all post first dose ADA responses less than (<) 9-fold over baseline titer levels; Treatment-boosted response - positive response in the assay post first dose, greater than or equal to (≥) 9-fold over baseline titer levels, when baseline results are positive; Treatment-emergent response - ADA positive response in the fasinumab ADA assay post first dose when baseline results = negative or missing.
Time Frame: Baseline up to week 72
Population: The ADA analysis set for the long-term safety population included all participants who received any study drug (SAF-LTS) and had at least 1 non-missing ADA result following the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W | Fasinumab 6 mg SC Q4W | Fasinumab 9 mg SC Q4W
Number analyzed (Participants) | 1153 | 911 | 929 | 208 | 1603 | 111 | 105
Participants
  ADA Negative Status | 1115 | 885 | 907 | 200 | 1547 | 108 | 104
  Pre-existing Immunoreactivity | 22 | 16 | 12 | 6 | 37 | 2 | 1
  Treatment-Boosted Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-Emergent Response | 16 | 10 | 10 | 2 | 19 | 1 | 0

13. Primary Outcome: Change From Baseline to Week 16 in the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Pain Subscale Score
Description: The WOMAC index is comprised of 24 parameters grouped in 3 subscales (pain-5 questions, physical function -17 questions and stiffness - 2 questions), with 0-10 grading of each question. The scores for each subscale are summed up, divided by number of questions, and each subscale is reported using Numerical Rating Scale score of 0-10. In addition to subscales, a total score is provided as the sum of normalized subscale scores divided by three, and reported using a Numerical Rating Scale score of 0-10. Higher scores indicate worse pain, stiffness and functional limitations.
Time Frame: Baseline to Week 16
Population: The full analysis set for the efficacy substudy (FAS-Substudy) included all randomized participants in the efficacy substudy. Here, Number of Participants Analyzed = Number of participants within a specified category.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W
Number analyzed (Participants) | 176 | 181 | 190 | 176 | 179
Score on a Scale | -1.55 (0.178) | -2.28 (0.175) | -2.77 (0.171) | -2.78 (0.174) | -2.59 (0.174)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 1 mg SC Q8W; Test type: Superiority; p = 0.0010, Mixed Models Analysis; Least Squares Mean = -0.73, 95% CI 2-sided [-1.159 to -0.293], Standard Error of Mean 0.221
Statistical Analysis 2: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean = -1.22, 95% CI 2-sided [-1.646 to -0.793], Standard Error of Mean 0.217
Statistical Analysis 3: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 3 mg SC Q4W; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean = -1.23, 95% CI 2-sided [-1.664 to -0.793], Standard Error of Mean 0.222
Statistical Analysis 4: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 6 mg SC Q8W; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean = -1.04, 95% CI 2-sided [-1.477 to -0.606], Standard Error of Mean 0.222

14. Primary Outcome: Change From Baseline to Week 16 in WOMAC Physical Function Subscale Score
Description: as for outcome 13
Time Frame: Baseline to Week 16
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W
Number analyzed (Participants) | 175 | 181 | 188 | 174 | 177
Score on a Scale | -1.35 (0.177) | -2.09 (0.175) | -2.55 (0.173) | -2.61 (0.177) | -2.48 (0.177)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 1 mg SC Q8W; Test type: Superiority; p = 0.0007, Mixed Models Analysis; Least Squares Mean = -0.74, 95% CI 2-sided [-1.163 to -0.309], Standard Error of Mean 0.218
Statistical Analysis 2: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean = -1.20, 95% CI 2-sided [-1.624 to -0.768], Standard Error of Mean 0.218
Statistical Analysis 3: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 3 mg SC Q4W; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean = -1.26, 95% CI 2-sided [-1.698 to -0.822], Standard Error of Mean 0.223
Statistical Analysis 4: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 6 mg SC Q8W; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean = -1.13, 95% CI 2-sided [-1.564 to -0.695], Standard Error of Mean 0.222

15. Secondary Outcome: Change From Baseline to Week 16 in Patient Global Assessment (PGA) Score of Osteoarthritis
Description: The PGA of OA is a patient-rated assessment of current disease state on a 5-point Likert scale (1 = very good; 2 = good; 3 = fair; 4 = poor; and 5 = very poor).
Time Frame: Baseline to Week 16
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W
Number analyzed (Participants) | 181 | 183 | 193 | 177 | 180
Score on a Scale | -0.66 (0.070) | -0.87 (0.071) | -0.93 (0.069) | -0.99 (0.071) | -0.96 (0.072)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 1 mg SC Q8W; Test type: Superiority; p = 0.0230, Mixed Models Analysis; Least Squares Mean = -0.20, 95% CI 2-sided [-0.380 to -0.028], Standard Error of Mean 0.090
Statistical Analysis 2: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.0025, Mixed Models Analysis; Least Squares Mean = -0.27, 95% CI 2-sided [-0.437 to -0.093], Standard Error of Mean 0.088
Statistical Analysis 3: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 3 mg SC Q4W; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Least Squares Mean = -0.32, 95% CI 2-sided [-0.496 to -0.145], Standard Error of Mean 0.090
Statistical Analysis 4: Comparison: Fasinumab-matching Placebo Q4W/Q8W vs Fasinumab 6 mg SC Q8W; Test type: Superiority; p = 0.0010, Mixed Models Analysis; Least Squares Mean = -0.29, 95% CI 2-sided [-0.466 to -0.118], Standard Error of Mean 0.089

16. Secondary Outcome: Number of Participants With ≥30% Reduction From Baseline to Week 16 in the WOMAC Pain Subscale Score
Description: The WOMAC index is comprised of 24 parameters grouped in 3 subscales (pain-5 questions, physical function -17 questions and stiffness - 2 questions), with 0-10 grading of each question. The scores for each subscale are summed up, divided by number of questions, and each subscale is reported using Numerical Rating Scale score of 0-10. In addition to subscales, a total score is provided as the sum of normalized subscale scores divided by three, and reported using a Numerical Rating Scale score of 0-10. Higher scores indicate worse pain, stiffness and functional limitations. Participants who achieved a response, where response was defined as an improvement by ≥30% in WOMAC pain subscale score
Time Frame: Baseline to Week 16
Population: The full analysis set for the efficacy substudy (FAS-Substudy) included all randomized participants in the efficacy substudy. Here, Number of Participants Analyzed = Number of participants within a specified category. Participants with missing data are considered as a non-response.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3 mg SC Q4W | Fasinumab 6 mg SC Q8W
Number analyzed (Participants) | 214 | 215 | 217 | 214 | 214
Participants | 76 | 108 | 126 | 118 | 114

ADVERSE EVENTS:
Time Frame: From time of randomization to end of post follow-up period (Week 100)
Groups:
- Fasinumab 1mg SC Q8W: Participants received fasinumab 1 mg SC injection, Q8W from day 1 up to 52 weeks.
- Fasinumab 1mg SC Q4W: Participants received fasinumab 1 mg SC injection Q4W from day 1 up to 52 weeks.
- Fasinumab 3mg SC Q4W: Participants received fasinumab 3 mg SC injection, Q4W from day 1 up to 52 weeks.
- Fasinumab 6mg SC Q8W: Participants received fasinumab 6 mg SC injection, Q8W from day 1 up to 52 weeks.
- Fasinumab 6mg SC Q4W: Participants received fasinumab 6 mg SC injection Q4W from day 1 up to 37 weeks of 52-week treatment period.
- Fasinumab 9mg SC Q4W: Participants received fasinumab 9 mg SC injection, Q4W from day 1 up to 37 weeks of 52-week treatment period.
Arm/Group | Fasinumab-matching Placebo Q4W/Q8W | Fasinumab 1mg SC Q8W | Fasinumab 1mg SC Q4W | Fasinumab 3mg SC Q4W | Fasinumab 6mg SC Q8W | Fasinumab 6mg SC Q4W | Fasinumab 9mg SC Q4W
All-Cause Mortality (participants affected / at risk) | 9/1257 | 5/966 | 8/974 | 0/214 | 12/1677 | 1/116 | 0/115
Serious Adverse Events (participants affected / at risk) | 183/1257 | 146/966 | 186/974 | 51/214 | 441/1677 | 29/116 | 26/115
Other Adverse Events (participants affected / at risk) | 988/1257 | 793/966 | 817/974 | 181/214 | 1447/1677 | 95/116 | 88/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasinumab-matching Placebo Q4W/Q8W (N=1257) | Fasinumab 1mg SC Q8W (N=966) | Fasinumab 1mg SC Q4W (N=974) | Fasinumab 3mg SC Q4W (N=214) | Fasinumab 6mg SC Q8W (N=1677) | Fasinumab 6mg SC Q4W (N=116) | Fasinumab 9mg SC Q4W (N=115)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular ataxia (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Terminal ileitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (18) | 16 (18) | 23 (25) | 5 (5) | 57 (62) | 3 (3) | 2 (2)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (14) | 11 (12) | 18 (19) | 8 (9) | 43 (44) | 4 (4) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (9) | 23 (23) | 27 (31) | 10 (11) | 157 (200) | 8 (10) | 6 (7)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 10 (10) | 0 (0) | 0 (0)
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 21 (21) | 2 (3) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Auditory nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 2 (3)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fistula (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial spasm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device loosening (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 9 (9) | 8 (8) | 9 (10) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 14 (15) | 14 (14) | 14 (14) | 5 (5) | 30 (33) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammatory carcinoma of breast stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axonal neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgic amyotrophy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Giant cell arteritis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diagnostic procedure (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Borderline glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Maculopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Idiopathic angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasinumab-matching Placebo Q4W/Q8W (N=1257) | Fasinumab 1mg SC Q8W (N=966) | Fasinumab 1mg SC Q4W (N=974) | Fasinumab 3mg SC Q4W (N=214) | Fasinumab 6mg SC Q8W (N=1677) | Fasinumab 6mg SC Q4W (N=116) | Fasinumab 9mg SC Q4W (N=115)
Arthralgia (Musculoskeletal and connective tissue disorders) | 413 (771) | 347 (636) | 350 (633) | 69 (109) | 710 (1358) | 53 (115) | 45 (82)
Back pain (Musculoskeletal and connective tissue disorders) | 204 (363) | 207 (336) | 185 (301) | 30 (37) | 283 (519) | 14 (24) | 13 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 113 (151) | 114 (144) | 124 (181) | 16 (31) | 151 (215) | 20 (29) | 12 (42)
Myalgia (Musculoskeletal and connective tissue disorders) | 77 (100) | 60 (81) | 58 (77) | 11 (11) | 101 (127) | 7 (7) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 74 (101) | 60 (87) | 75 (101) | 30 (38) | 116 (150) | 7 (10) | 6 (7)
Joint swelling (Musculoskeletal and connective tissue disorders) | 37 (43) | 32 (33) | 35 (38) | 15 (17) | 143 (183) | 4 (6) | 10 (12)
Headache (Nervous system disorders) | 395 (1445) | 370 (948) | 418 (1081) | 76 (158) | 554 (1833) | 34 (124) | 30 (73)
Paraesthesia (Nervous system disorders) | 42 (54) | 54 (66) | 76 (95) | 13 (18) | 144 (169) | 6 (6) | 9 (10)
Hypoaesthesia (Nervous system disorders) | 35 (43) | 25 (32) | 27 (31) | 11 (14) | 100 (130) | 5 (6) | 8 (12)
Carpal tunnel syndrome (Nervous system disorders) | 28 (31) | 42 (49) | 49 (58) | 17 (19) | 116 (135) | 11 (12) | 10 (16)
Nasopharyngitis (Infections and infestations) | 184 (233) | 189 (289) | 211 (304) | 43 (55) | 224 (279) | 12 (12) | 18 (21)
Upper respiratory tract infection (Infections and infestations) | 142 (198) | 82 (103) | 89 (113) | 17 (17) | 220 (297) | 15 (18) | 10 (13)
Urinary tract infection (Infections and infestations) | 126 (171) | 84 (107) | 125 (161) | 21 (26) | 160 (217) | 9 (11) | 6 (9)
Influenza (Infections and infestations) | 69 (88) | 54 (59) | 59 (66) | 10 (10) | 103 (119) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 110 (159) | 91 (148) | 118 (176) | 11 (14) | 118 (188) | 5 (5) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 58 (67) | 55 (67) | 46 (61) | 10 (10) | 81 (88) | 13 (19) | 4 (8)
Peripheral swelling (General disorders) | 16 (20) | 11 (11) | 20 (23) | 5 (6) | 81 (97) | 3 (3) | 11 (11)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 26 (27) | 51 (55) | 70 (73) | 17 (19) | 170 (214) | 11 (11) | 8 (10)
Dizziness (Nervous system disorders) | 61 (75) | 45 (49) | 48 (61) | 7 (7) | 94 (109) | 10 (17) | 7 (10)
Sciatica (Nervous system disorders) | 24 (30) | 27 (31) | 33 (34) | 10 (10) | 75 (88) | 6 (7) | 3 (3)
Bronchitis (Infections and infestations) | 53 (55) | 34 (35) | 33 (36) | 4 (4) | 73 (79) | 7 (7) | 3 (4)
Sinusitis (Infections and infestations) | 31 (34) | 23 (27) | 20 (22) | 5 (5) | 71 (80) | 7 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 37 (41) | 26 (27) | 22 (24) | 2 (3) | 45 (48) | 5 (6) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 54 (62) | 48 (54) | 56 (62) | 9 (10) | 65 (79) | 5 (7) | 5 (6)
Contusion (Injury, poisoning and procedural complications) | 34 (42) | 35 (48) | 36 (48) | 7 (7) | 62 (70) | 2 (2) | 8 (9)
Hypertension (Vascular disorders) | 54 (56) | 54 (59) | 47 (51) | 7 (8) | 80 (84) | 2 (2) | 4 (4)
Oedema peripheral (General disorders) | 32 (38) | 26 (29) | 24 (25) | 9 (9) | 95 (112) | 11 (11) | 5 (5)
Limb injury (Injury, poisoning and procedural complications) | 19 (19) | 21 (28) | 30 (31) | 3 (4) | 37 (41) | 5 (5) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT02683239/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT02683239/SAP_001.pdf